CLINICAL TRIAL: NCT07088315
Title: Clinical Effects of TECAR Therapy in the Conservative Management of Lipedema: A Randomized Controlled Trial
Brief Title: Effects of TECAR Therapy in Lipedema Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Oznur Uzun, MD, Deputy Chief of Physical Medicine and Rehabilitation Hospital, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TABED 1-24-324
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Lipedema
Keywords: Lipedema; TECAR Therapy; Pain Management; Quality of Life
MeSH Terms: conditions — Lipedema; Agnosia | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group receiving exercise and compression (Active Comparator): All participants were provided with individually fitted compression garments (either pantyhose-type or thigh-high models, in class I [18-21 mmHg] or class II [23-32mmHg] depending on symptom severity and tolerance), and were instructed to wear them during waking hours for a minimum of 8 hours per day. Adherence to garment usage was monitored through patient diaries and reinforced at follow-up visits.
  Additionally, all patients were advised to engage in a structured walking program, consisting of moderate-intensity walking (perceived exertion level 11-13 on the Borg scale), for at least 20 minutes per session, three times per week.
  Interventions: Other: compression; Other: Exercise
- The treatment group receiving exercise and compression plus TECAR Therapy (Experimental): TECAR therapy was applied to the lower limbs of patients diagnosed with lipedema using the BTL-6000 TR-Therapy PRO device (BTL, Turkiye). All treatment sessions were performed by a physiotherapist with specific experience in TECAR therapy. The device operated at a frequency of approximately 500 kHz and employed three types of electrodes: active, neutral, and static application electrodes. Two types of active electrodes -capacitive and resistive- were utilized and applied directly to the treatment area. The neutral electrode, serving as a reference point, was placed in proximity to the target region to ensure effective energy transfer.
  Interventions: Device: TECAR therapy; Other: compression; Other: Exercise

INTERVENTIONS:
Device: TECAR therapy — TECAR therapy was applied to the lower limbs of patients diagnosed with lipedema using the BTL-6000 TR-Therapy PRO device (BTL, Turkiye). All treatment sessions were performed by a physiotherapist with specific experience in TECAR therapy. The device operated at a frequency of approximately 500 kHz and employed three types of electrodes: active, neutral, and static application electrodes. Two types of active electrodes -capacitive and resistive- were utilized and applied directly to the treatment area. The neutral electrode, serving as a reference point, was placed in proximity to the target region to ensure effective energy transfer.
  Arms: The treatment group receiving exercise and compression plus TECAR Therapy
Other: compression — All participants were provided with individually fitted compression garments (either pantyhose-type or thigh-high models, in class I [18-21 mmHg] or class II [23-32mmHg] depending on symptom severity and tolerance), and were instructed to wear them during waking hours for a minimum of 8 hours per day. Adherence to garment usage was monitored through patient diaries and reinforced at follow-up visits.
Other: Exercise — All patients were advised to engage in a structured walking program, consisting of moderate-intensity walking (perceived exertion level 11-13 on the Borg scale), for at least 20 minutes per session, three times per week.

SUMMARY:
The physicians wanted to show the efficacy of a physical therapy device, Transfer Energy Capacitive and Resistive (TECAR) therapy, in women with lipedema which is an abnormal fat buildup on both sides of lower body. They focused on lower limb circumference, pain, functional capacity, and quality of life.

DETAILED DESCRIPTION:
This study aimed to evaluate the clinical efficacy of Transfer Energy Capacitive and Resistive (TECAR) therapy in women with Stage 2 lipedema, focusing on limb circumference, pain, functional status, and quality of life.

A prospective, randomized controlled trial was conducted with 30 female patients diagnosed with Stage 2 lipedema. Participants were randomized to a TECAR therapy group (n=15) or a control group (n=15). Both groups received compression garments and a structured exercise program; the TECAR group additionally underwent six TECAR sessions over three weeks. Outcomes included lower limb circumference, Visual Analog Scale (VAS) for pain, Lower Extremity Functional Scale (LEFS), and Lymphedema Quality of Life Questionnaire-Leg (LYMQOL-Leg), assessed at baseline and at one and three months post-treatment.

TECAR therapy resulted in greater reductions in lower limb circumference compared to standard care, with sustained improvement in the supramalleolar region at three months (p<0.05). A significant short-term reduction in pain was observed at one month (p = 0.003) only in the TECAR group, but this effect was not maintained at three months (p > 0.05). Functional scores trended toward improvement without reaching significance (p=0.058). The overall quality of life score improved significantly in the TECAR group (p=0.002), although individual LYMQOL subdomains including function, appearance, mood, or symptoms did not reach statistical significance (p > 0.05).

As an adjunct to standard care, TECAR therapy appears to reduce pain and limb volume and enhance overall quality of life in Stage 2 lipedema. Further long-term studies are needed to confirm these findings.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 60 years
* Clinical diagnosis of Stage 2 lipedema (types 1-3)
* Body mass index (BMI) which is less than 35

Exclusion Criteria:

* Deterioration in general condition,
* Presence of open wounds or sensory deficits in the area of application,
* Active infections,
* Malignancy,
* Autoimmune or systemic inflammatory diseases (e.g., rheumatoid arthritis or systemic lupus erythematosus),
* Severe cognitive impairment,
* Uncontrolled chronic systemic disease,
* History of physiotherapy or regular non-steroidal anti-inflammatory drug (NSAID) use within the last six months
* Concomitant lymphedema or venous insufficiency.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Circumference measurements | Clinical assessments were conducted at baseline, as well as at 1 and 3 months following the treatment.
  Circumference measurements were performed using a standard non-elastic tape measure at three anatomically defined landmarks: the mid-thigh, identified as the midpoint between the iliac crest and the lower border of the patella, the pretibial region, defined as the midpoint between the anterior tibial tuberosity and the medial malleolus and supramalleolar region. These regions were selected for their clinical relevance in lipedema and their high reproducibility in anthropometric assessments. To enhance measurement reliability, each site was measured three times consecutively, and the mean value was used for analysis. All measurements were conducted with the patient in a relaxed standing position by the same examiner to minimize inter-observer variability.
visual analogue scale (VAS) | Clinical assessments were conducted at baseline, as well as at 1 and 3 months following the treatment.
  Pain intensity was evaluated using the Visual Analog Scale (VAS), a 10-cm horizontal line representing a continuum of pain experience, where 0 indicates "no pain" and 10 denotes the "worst imaginable pain". Participants were asked to mark the point that best reflected their pain perception at each evaluation time point.
The Lower Extremity Functional Scale (LEFS) | Clinical assessments were conducted at baseline, as well as at 1 and 3 months following the treatment.
  Functional status was evaluated using the LEFS, a widely validated, patient-reported outcome measure specifically designed to assess lower extremity functional impairment. The LEFS consists of 20 items, each addressing a different daily or recreational activity involving the legs, such as walking, climbing stairs, squatting, or running. Participants rated the level of difficulty they experienced performing each activity on a 5-point Likert scale, ranging from 0 (extreme difficulty or unable to perform) to 4 (no difficulty).The total score ranges from 0 to 80, with higher scores reflecting greater functional capacity and less disability
The Lymphedema Quality of Life Questionnaire for the Leg (LYMQOL-Leg) | Clinical assessments were conducted at baseline, as well as at 1 and 3 months following the treatment.
  Quality of life was assessed using LYMQOL-Leg, a disease-specific instrument originally designed to evaluate health-related quality of life in patients with lower limb lymphedema. The questionnaire includes 24 items grouped into four distinct domains: function (activities of daily living and physical capacity), appearance (self-perception of leg aesthetics), mood (emotional and psychological well-being), and symptoms (such as heaviness, swelling, and pain). Each item is scored on a Likert scale from 1 to 4, with lower scores indicating greater impairment. In addition to domain scores, the LYMQOL includes a global quality of life score (rated on a scale from 0 to 10), where higher values reflect better overall quality of life [23, 24]. Although originally developed for lymphedema, LYMQOL has been effectively applied in lipedema studies due to symptom overlap.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Physical Medicine and Rehabilitation Hospital, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD can be shared upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: The doctors specialized in physical medicine and rehabilitation may reach principal investigator through email

REFERENCES:
- [Background] Atan T, Bahar-Ozdemir Y. The Effects of Complete Decongestive Therapy or Intermittent Pneumatic Compression Therapy or Exercise Only in the Treatment of Severe Lipedema: A Randomized Controlled Trial. Lymphat Res Biol. 2021 Feb;19(1):86-95. doi: 10.1089/lrb.2020.0019. Epub 2020 Dec 9. PMID 33297826
- [Background] Kruppa P, Gohlke S, Lapinski K, Garcia-Carrizo F, Soultoukis GA, Infanger M, Schulz TJ, Ghods M. Lipedema stage affects adipocyte hypertrophy, subcutaneous adipose tissue inflammation and interstitial fibrosis. Front Immunol. 2023 Jul 28;14:1223264. doi: 10.3389/fimmu.2023.1223264. eCollection 2023. PMID 37575263
- [Background] Kruppa P, Georgiou I, Biermann N, Prantl L, Klein-Weigel P, Ghods M. Lipedema-Pathogenesis, Diagnosis, and Treatment Options. Dtsch Arztebl Int. 2020 Jun 1;117(22-23):396-403. doi: 10.3238/arztebl.2020.0396. PMID 32762835
- [Background] Faerber G, Cornely M, Daubert C, Erbacher G, Fink J, Hirsch T, Mendoza E, Miller A, Rabe E, Rapprich S, Reich-Schupke S, Stucker M, Brenner E. S2k guideline lipedema. J Dtsch Dermatol Ges. 2024 Sep;22(9):1303-1315. doi: 10.1111/ddg.15513. Epub 2024 Aug 27. PMID 39188170